CLINICAL TRIAL: NCT02137668
Title: The Human Gastrointestinal Tract Microbiota in the Setting of Treating Primary Sclerosing Cholangitis and Biliary Atresia With Vancomycin
Brief Title: Treating Primary Sclerosing Cholangitis and Biliary Atresia With Vancomycin
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sacramento Pediatric Gastroenterology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Davies 1
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Primary Sclerosing Cholangitis; Biliary Atresia
MeSH Terms: conditions — Cholangitis, Sclerosing; Biliary Atresia | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral Vancomycin (Experimental): Every participant with PSC or BA will received the same Arm of Oral Vancomycin
  Interventions: Drug: Oral Vancomycin

INTERVENTIONS:
Drug: Oral Vancomycin — Oral Vancomycin is given to PSC or BA participants
  Other Names: ANI

SUMMARY:
The purpose of this study is twofold. First, is to determine whether vancomycin is effective in the early treatment of Biliary Atresia (BA) and Primary Sclerosing Cholangitis (PSC), and if so, by what mechanism. Secondly, to characterize human intestinal microbial communities and their interactions with the host.

DETAILED DESCRIPTION:
Investigators hope to learn to characterize human intestinal microbial communities (microbiome: the collection or collectivity of microorganisms) using molecular methods, examine the mechanisms of interaction between host and microbiome using genomic approaches, and determine how the microbiome both preserves local health and promotes pathology. Investigation will focus on primary sclerosing cholangitis, biliary atresia, as well as states of health. The composition of the associated microbiome will be assessed based on ribosomal DNA and RNA sequences, and attention will be given to richness (diversity), evenness (relative abundance), and variation with respect to time, person, and anatomic niche. Host response at the adjacent mucosal surface will be assessed based on genome-wide gene expression patterns. In addition, changes in the metabolites of the blood will be analyzed.

To see if the antibiotic vancomycin, when used for the early treatment of Biliary Atresia (BA) and Primary Sclerosing Cholangitis (PSC) is effective treatment for these diseases. Investigators hope to learn what effect Vancomycin has on the bacteria that are present in stool, body fluid or intestinal tissue on someone who has BA and PSC and if so by what mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Persons who have primary sclerosing cholangitis, biliary atresia, a chronic intestinal disorder or who are undergoing upper or lower endoscopy.
* Persons who have primary sclerosing cholangitis or biliary atresia who are good candidates for vancomycin therapy.

Exclusion Criteria:

* Patients that have taken antibiotics and/or immunomodulators within the last 3 months will be excluded as this will alter the original bacterial flora.
* Females who are pregnant may not participate.

Ages: 2 Weeks to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-07; Primary Completion 2018-05 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Determine the benefit of oral vancomycin therapy for Primary Sclerosing Cholangitis and Biliary Atresia | 3 months
  Blood tests, imaging studies and/or liver biopsy changes before and while on oral vancomycin will determine the benefit of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yinka Davies, M.D., Principal Investigator — Sacramento Pediatric Gastroenterology
Locations (1):
- Sacramento Pediatric Gastroenterology, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected throughout study and will be shared via publications when available at certain time points.